CLINICAL TRIAL: NCT04837833
Title: Machine Learning Approach to Sonographic Assessment of Tumor Volumes for Response Assessment in Patients With Pancreas or Gastrointestinal Adenocarcinoma: A Pilot Study
Brief Title: An Ultrasound Imaging Technique to Measure Tumors in People With Pancreatic Ductal Adenocarcinoma (PDAC) or Gastrointestinal (GI) Adenocarcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-138
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pancreas Cancer; Gastrointestinal Adenocarcinoma
Keywords: Sonographic Assessment; Tumor Volumes for Response; 21-138
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- research ultrasound (rUS1) (Experimental): Participants will undergo research ultrasound (rUS1) within three days of their routine contrast enhanced CT scan (CECT). A subset of participants (up to 10) will undergo a second research US (rUS2) at 3-4 weeks after rUS1 and at least one month prior to the next planned clinical CECT.
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — Participants will undergo research ultrasound (rUS1) within three days of their routine CECT scan. A subset of participants (up to 10) will undergo a second research US (rUS2) at 3-4 weeks after rUS1 and at least one month prior to the next planned clinical CECT

SUMMARY:
The purpose of this study is to see if ultrasound images that are analyzed by a special computer program can be used to measure the size of PDAC tumors in the liver as accurately as CT scans that involve contrast material (also called contrast-enhanced CT scans). All participants in this study will have pancreatic ductal adenocarcinoma (PDAC) that has spread (metastasized) to the liver, and all participants will be scheduled for a routine CT scan that will measure their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 18 years of age or older
* Confirmed diagnosis of PDAC or GI tract adenocarcinoma metastatic to liver
* Scheduled for imaging with contrast enhanced CT

Exclusion Criteria:

* Inability to tolerate intravenous contrast medium
* All liver metastases ≤ 10 mm in maximal diameter on the contrast enhanced CT used for comparison to the planned research ultrasound
* Multiple confluent liver metastases or tumor burden > 50% of the liver as estimated by a radiologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
measurement differences between ultrasound tumor volumes | 1 year
  Measure the range of volumetric changes of liver metastases observed between rUS1 and rUS2. We will correlate the rate (%) of tumor volumetric change between the rUS1 and rUS2 to the rate of change between the two CECT.

CONTACTS AND LOCATIONS:
Overall Officials: Kinh Gian Do, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm